CLINICAL TRIAL: NCT01471912
Title: Asymmetric Elongation of Foveal Tissue After Macular Hole Surgery and Its Impact on Metamorphopsia
Brief Title: Elongation of Foveal Tissue After Macular Hole Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-10-003
Record Dates: First submitted 2011-11-06; First posted 2011-11-16 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Macular Holes
Keywords: Macular Holes; spectral domain optical coherence tomography; elongation of foveal tissue; M-score
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: pars plana vitrectomy and fluid gas exchange — A three-port standard pars plana vitrectomy was performed by a single surgeon using a 23-gauge vitrectomy system, either Associate®(Dutch Ophthalmic Research Center. Inc., Zuidland, The Netherlands) or Accurus®(Alcon Laboratories Inc., Fort Worth, USA), with one step scleral tunnel incision. In all cases, the peeling of the internal limiting membrane, approximately 1 disc diameter area from center of MH was conducted without assistance of dyes followed by complete fluid-gas exchange using 25% sulfur hexafluoride gas. Combined cataract surgery was performed in patients with visually significant cataracts or with incipient cataract in the subjects older than 60 years. All patients were instructed to maintain a face-down position for at least 7 days postoperatively.

SUMMARY:
In our experience, elongation of foveal tissue after macular hole surgery which was undetectable by conventional time-domain optical coherence tomography was often observed on spectral-domain optical coherence tomography images. Elongation of tissues inevitably induces some degree of disorganization of tissue microstructure.

The purpose of the present study was to evaluate elongation profile of foveal tissue after macular hole surgery and to investigate its impact on visual acuity and metamorphopsia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with idiopathic macular hole

Exclusion Criteria:

* traumatic macular hole
* evidence of ocular inflammation, diabetic retinopathy, hypertensive retinopathy, and retinal vasculitis, media opacity that would influence visual acuity or preclude acquisition of clear spectral domain optical coherence tomography images
* presence of cataract judged to affect visual function, -6.0 diopters or more of spherical equivalent, prominent staphyloma
* history of intraocular surgery other than uncomplicated cataract surgery, other ocular diseases that may influence the macular microstructure or visual function
* patients with indistinct intraretinal structure on spectral domain optical coherence tomography images

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Changes in the inter-outer plexiform layer distance | first postoperative visit, 1 month, 2 months, and 6 months after macular hole surgery
  the spectral domain optical coherence tomography scannings were performed at first postoperative visit, 1 month, 2 months, and 6 months after macular hole surgery. The inter-outer plexiform layer distance was measured based on optical coherence tomography images at defined time points
Changes in best-corrected visual acuity | first postoperative visit, 2 months, and 6 months after macular hole surgery
  Best-corrected visual acuity was measured using early treatment diabetic retinopathy study chart at defined time points
Changes in degree of metamorphopsia | first postoperative visit, 2 months, and 6 months after macular hole surgery
  The degree of metamorphopsia was measured using Metamorphopsia-chart at defined time points
Degree of percent asymmetric elongation on the same plane | at 6 months postoperative
  The horizontal percent asymmetry was calculated as (nasal distance - temporal distance)/(nasal distance + temporal distance). The vertical percent asymmetry was also calculated as (superior distance - inferior distance)/ (superior distance + inferior distance.
Degree of horizontal-vertical percent asymmetry | at 6 months postoperative
  The percent asymmetry was calculated as (horizontal inter-outer plexiform layer distance - vertical inter-outer plexiform layer distance)/(horizontal inter-outer plexiform layer distance + vertical inter-outer plexiform layer distance).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea